CLINICAL TRIAL: NCT03266406
Title: Effect of Hyaluronidase on Intraocular Pressure After Retrobulbar Anaesthesia During Cataract Surgery
Brief Title: Effect of Hyaluronidase on Intraocular Pressure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Eman Yassin Ahmed, Principal Investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: effect of hyaluronidase on IOP
Record Dates: First submitted 2017-08-28; First posted 2017-08-30 (Actual); Last update posted 2017-08-30 (Actual); Status verified 2017-08

CONDITIONS: Intraocular Pressure Low
MeSH Terms: conditions — Ocular Hypotension | interventions — Hyaluronoglucosaminidase

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Effect of hyaluronidase on IOP (Experimental)
  Interventions: Drug: Hyaluronidase

INTERVENTIONS:
Drug: Hyaluronidase — 4ml of retrobulbar LA with addition of 15IU/ml hyaluronidase to 2% lidocaine

SUMMARY:
The aim of this study is to evaluate effect of retrobulbar local anaesthesia after addition of hyaluronidase on IOP during cataract surgery

ELIGIBILITY:
Inclusion Criteria:

* 1-Patients above the age of 50 years. 2-Patients with age related cataract. 3-Normal IOP.

Exclusion Criteria:

* 1History of trauma. 2-Patients with glaucoma. 3-Previous ocular surgery. 4-Patients with other ocular pathology. 5-Uncontrolled diabetes or hypertension. 6-hypersensitivity to lignocaine. 7-Uncooperative or epileptic patients.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-09 (Estimated); Primary Completion 2018-09 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
reduction in IOP | within 10minutes
  reduction of complications of high IOP during surgery